CLINICAL TRIAL: NCT02786108
Title: Bariatric Arterial Embolization for Morbid Obesity
Acronym: BAEMO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Professor of Radiology & Chair,Department of Radiology, Zhongda Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015ZDSYLL068.0
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Morbid Obesity
Keywords: left gastric artery; embolization; obesity
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Diet, Healthy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- left gastric artery embolization (Experimental): Patients undergoing left gastric artery embolization
  Interventions: Procedure: left gastric artery embolization
- healthy diet and exercise (Active Comparator): Patients undergoing healthy diet and exercise
  Interventions: Behavioral: healthy diet and exercise

INTERVENTIONS:
Procedure: left gastric artery embolization
  Arms: left gastric artery embolization
Behavioral: healthy diet and exercise
  Arms: healthy diet and exercise

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of left gastric artery embolization(bariatric arterial embolization) for morbid obesity. When the target vessel is blocked, some of the body's signals for feeling hungry will be suppressed and lead to weight loss.

Although there are many ways to treat morbid obesity, surgery is currently the only effective method to be confirmed. But surgical treatment is likely to carry a high risk of treatment-related complications, such as fistula or intestinal obstruction, etc. This study is designed to help treat obesity using a method of transvascular interventional therapy, which is minimally invasive and non-surgical.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) >30.
2. No history of gastrointestinal surgery.
3. Willing, able and mentally competent to provide written informed consent.
4. Suitable for protocol therapy as determined by the interventional radiology Investigator.
5. Adequate hematological, hepatic and renal function as follows:

   Hematological Neutrophils > 1.5 x 109/L Platelets > 100 x 109/L INR <1.5 Hepatic Bilirubin ≤ 2.0 mg/dL Albumin ≥ 2.5 g/L Renal Estimated GFR > 60ml/min.1.73m2
6. Aged between18 and 65 years old.
7. More than one year's follow-up can be obtained reliably

Exclusion Criteria:

1. Prior history of gastric pancreatic, hepatic, and/or splenic surgery
2. Prior embolization to the stomach, spleen or liver
3. Prior or current history of peptic ulcer disease
4. Significant risk factors for peptic ulcer disease including daily NSAID use and smoking.
5. Portal venous hypertension or cirrhosis
6. Less than 18 years or older than 65 years of age
7. Known aortic pathology such as aneurysm or dissection renal insufficiency as evidenced by an estimated glomerular filtration rate of < 60 milliliters per minute an estimated glomerular filtration rate of < 60 milliliters per minute
8. Major comorbidity such as cancer, significant cardiovascular disease, or peripheral arterial disease
9. Pregnant or intend to become pregnant within one year Known history of allergy to iodinated contrast media
10. Patients with certain psychiatric disorders such as schizophrenia, borderline personality disorder, and uncontrolled depression, and mental/cognitive impairment that limits the individual's ability to understand the proposed therapy.
11. Patients currently taking or requiring chronic use of NSAID or steroid medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-10 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | Baseline, post-op 1 month, 3 months, 6 months,9 months,12 months
  Unit of Measure: Percentage of excess weight loss [%EWL]. The body weight will be measured within 2-4h after breakfast.

SECONDARY OUTCOMES:
Blood pressure | Baseline, post-op 1 month, 3 months, 6 months,9 months,12 months
  The brachial artery blood pressure will be measured in the early hours of the morning and under the quiet situation. Unit of Measure: mmHg.
Lipid Profile | Baseline, post-op 1 month, 3 months, 6 months,9 months,12 months
  Blood cholesterol levels, triglyceride levels and lipoprotein levels will be detected. Unit of Measure: mmol/L.
Number of Patients with Adverse Events | post-op 30 days
  Surgical complications and adverse events such as massive hemorrhage, femoral artery pseudoaneurysm, gastric mucosal ischemia and necrosis and gastric perforation, etc., will be documented.
Ghrelin levels | Baseline, post-op 1 month, 3 months, 6 months,9 months,12 months
  Unit of Measure: pg/mL. Detection of serum Ghrelin levels will be obtained using fasting blood in the morning.
Abdominal fat content | Baseline, post-op 1 month,6 months,12 months
  Abdominal fat content detected by MRI.
Leptin levels | Baseline, post-op 1 month, 3 months, 6 months,9 months,12 months
  Detection of serum Leptin levels will be obtained using fasting blood in the morning. Unit of Measure: pg/mL.
Results of Gastroendoscopic Examination | Baseline, post-op 1 week, post-op 1 month, 3 months, 6 months,9 months,12 months
  Photos and clinical reports will be analyzed.
Quality of Life Parameters Survey | 12 months
  N/A Utilizing SF-36/ pre and post procedure to determine the changes of quality in life; everyday activities.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-jun Teng, Ph.D,MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital,Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Bai ZB, Qin YL, Deng G, Zhao GF, Zhong BY, Teng GJ. Bariatric Embolization of the Left Gastric Arteries for the Treatment of Obesity: 9-Month Data in 5 Patients. Obes Surg. 2018 Apr;28(4):907-915. doi: 10.1007/s11695-017-2979-9. PMID 29063494